CLINICAL TRIAL: NCT00212459
Title: A Prospective Randomized Pilot Study on the Effect of Patient Counseling on Adolescent Hemophilia Patient Compliance With Bleeding Logs
Brief Title: The Effect of Patient Counseling on Adolescent Hemophilia Patient Compliance With Bleeding Logs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Donna DiMichele, MD, New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Bleeding Logs
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2008-05

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Bleeding logs; Factor Infusions
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients are contacted every two weeks after initial counseling to discuss completion of bleeding records.
  Interventions: Behavioral: Counseling
- 2 (Active Comparator): After the initial counseling with regards to bleeding records, there are no more contacts made with the control patients.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Counseling — Patients are contacted every two weeks after initial counseling to discuss the completion of bleeding records.
  Arms: 1
Behavioral: Control — No more contacts are made with control patients after the initial counseling session.
  Arms: 2

SUMMARY:
The study will see if counselling adolescents with severe or moderate Hemophilia A or B results in increased compliance in the maintenance of bleeding logs.

DETAILED DESCRIPTION:
The study will see if counselling adolescents with severe or moderate Hemophilia A or B results in increased compliance in the maintenance of bleeding logs.To do this subjects will be randomized into a control group and a group who will receive consistent counselling by a pharmacist about their bleeding logs.

The aims of the study are:

* To provide a new method of bleeding and treatment documentation in the home setting (logs) to adolescent subjects with Hemophilia A or B
* To counsel these subjects about adherence to their treatment regimen prescribed by physician and the importance of keeping accurate documentation of each bleeding episode and its treatment.
* To improve maintenance of logs, to allow for 1) assessment of bleeding frequency and treatment efficacy and 2) early detection of target joint bleeding and the potential need for prophylactic factor replacement.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 through 20
* Severe or moderate Hemophilia A or B
* Self-infusing or transitioning to self infusion in the home setting
* Already assigned responsibility of monitoring bleeding logs

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 12 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2005-05; Primary Completion 2006-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Study and control groups will be compared with respect to the % of bleeds reported to the HTC and % of recommended therapy recorded in bleeding logs after a 6 month period | 6 months

SECONDARY OUTCOMES:
Study and control groups will be compared with respect to time between initiation of target joint bleeding and the identification and treatment of such by HTC personnel | 6 months
Clotting factor consumption and the cost of therapy in each group will be compared | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Donna M DiMichele, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NY Presbyterian Hospital, New York, New York, United States